CLINICAL TRIAL: NCT00840086
Title: A Multi-centre, Open-label, Non-controlled Trial on Safety and Efficacy of N8 in Prevention and Treatment of Bleeds in Previously Treated Subjects With Haemophilia A. Sub-trial: Safety and Efficacy of N8 in Prevention and Treatment of Bleeding During Surgical Procedures in Subjects With Haemophilia A
Brief Title: Safety and Efficacy of Turoctocog Alfa in Haemophilia A Subjects
Acronym: guardian™1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3543; 2008-003960-20 (EudraCT Number); 101151 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFVIII (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Subjects will receive bleeding preventive treatment (home treatment with self-injection i.v.) with turoctocog alfa at a dose of 20-40 IU/kg body weight every second day or 20-50 IU/kg body weight three times per week at the investigator's discretion.

SUMMARY:
This trial is conducted in Asia, Europe, and North and South America. The trial consists of a main trial and a sub-trial. The main trial investigates safety and efficacy of turoctocog alfa (recombinant factor VIII, rFVIII (N8)) in haemophilia A subjects, while the sub-trial investigates safety and efficacy of turoctocog alfa in prevention and treatment of bleeding episodes during surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with the diagnosis of severe (FVIII less than or equal to 1%) haemophilia A from age 12 (except for Israel where the age limit will be 18 for the first 10 subjects recruited in the trial) to 56 years having a weight of 10 to 120 kg
* Documented history of at least 150 exposure days to any other FVIII products (prevention or treatment of bleeds)
* No history of FVIII inhibitors greater than or equal to 0.6 BU/mL. The inhibitor should be measured regularly for at least the last 8 years or since the first treatment of haemophilia A
* No detectable inhibitors to FVIII (greater than or equal to 0.6 BU/mL) (as assessed by a Central Laboratory at the time of screening)

Exclusion Criteria:

* Congenital or acquired coagulation disorders other than haemophilia A
* Creatinine levels 50% above normal level (as defined by central laboratory range)
* Known or suspected allergy to trial product (N8) or related products

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (59):
- United States (18):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Spokane, Washington
- Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Croatia (2):
  - Novo Nordisk Investigational Site, Split
  - Novo Nordisk Investigational Site, Zagreb
- Novo Nordisk Investigational Site, Copenhagen, Denmark
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (9):
  - Novo Nordisk Investigational Site, Hiroshima-shi, Hiroshima
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Saint Petersburg, Russia
- Serbia and Montenegro (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Nis
  - Novo Nordisk Investigational Site, Novi Sad
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit
  - Novo Nordisk Investigational Site, Samsun
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] Lentz SR, Misgav M, Ozelo M, Salek SZ, Veljkovic D, Recht M, Cerqueira M, Tiede A, Brand B, Mancuso ME, Seremetis S, Lindblom A, Martinowitz U. Results from a large multinational clinical trial (guardian1) using prophylactic treatment with turoctocog alfa in adolescent and adult patients with severe haemophilia A: safety and efficacy. Haemophilia. 2013 Sep;19(5):691-7. doi: 10.1111/hae.12159. Epub 2013 May 7. PMID 23647704
- [Result] Santagostino E, Lentz SR, Misgav M, Brand B, Chowdary P, Savic A, Kilinc Y, Amit Y, Amendola A, Solimeno LP, Saugstrup T, Matytsina I. Safety and efficacy of turoctocog alfa (NovoEight(R)) during surgery in patients with haemophilia A: results from the multinational guardian clinical trials. Haemophilia. 2015 Jan;21(1):34-40. doi: 10.1111/hae.12518. Epub 2014 Oct 2. PMID 25273984
- [Result] Ozelo M, Chowdary P, Regnault A, Busk AK. Impact of severe haemophilia A on patients' health status: results from the guardian() 1 clinical trial of turoctocog alfa (NovoEight((R)) ). Haemophilia. 2015 Jul;21(4):451-7. doi: 10.1111/hae.12617. Epub 2015 Feb 12. PMID 25677761
- [Result] Ozelo MC. Updates from guardian: a comprehensive registration programme. Eur J Haematol. 2015 Dec;95 Suppl 81:22-9. doi: 10.1111/ejh.12648. PMID 26679394
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited at 48 sites in 15 countries: Republic of Serbia (5), Turkey (5), Germany (4), Japan (8), the United Kingdom (3) and the United States of America (10). Two sites each in Brazil, Italy, Spain and Croatia. One site each in Switzerland, Taiwan, Israel, Malaysia and Russian Federation.
Groups:
- All Subjects Treated With Turoctocog Alfa: All subjects participating in the study (Part A + Part B + Part C).
Period: Overall Study
Arm/Group | All Subjects Treated With Turoctocog Alfa
Started | 150
Completed | 146
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 150
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic Or Latino | 25
  Not Hispanic Or Latino | 125
Region of Enrollment [Number; unit: participants]
  Brazil | 16
  Croatia | 11
  Germany | 10
  Israel | 12
  Italy | 7
  Japan | 9
  Malaysia | 5
  Russia | 5
  Serbia | 19
  Spain | 4
  Switzerland | 5
  Taiwan | 4
  Turkey | 11
  United Kingdom | 3
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: The Incidence Rate of FVIII Inhibitors (Greater Than or Equal to 0.6 Bethesda Units (BU))
Description: The incidence rate of FVIII inhibitors was calculated by including all patients with inhibitors in the nominator and including all patients with a minimum 50 exposure plus any patients with less than 50 exposures but with inhibitors in denominator.
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 188 days per subject.
Population: The safety analysis set includes all 150 subjects who received at least one dose of the investigational product. The analysis of the primary endpoint included all subjects with at least 50 exposure days and/or with inhibitors. A total of 148 subjects had 50 exposure days (EDs).
Measure: Number; unit: N with Inhibitors / N with ≥50 EDs
Arm/Group | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 148
N with Inhibitors / N with ≥50 EDs | 0

2. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Adverse event was defined as events occurring after administration of trial product. Severe AEs: considerable interference with subject's daily activities, unacceptable. Moderate AEs: Marked symptoms, moderate interference with the patient's daily activities. Mild AEs: No or transient symptoms, no interference with the patient's daily activities. Serious AEs: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalization, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 188 days per subject
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Number; unit: events
Groups:
- Total (Part A + Part B): Preventive treatment and treatment of bleeds: The doses were individualised based on the trough FVIII activity level. The doses could be adjusted by the investigator. The dose level chosen was 20-40 IU/kg every second day or 20-50 IU/kg three times per week (Part A + Part B). Subjects previously treated with turoctocog alpha were included in Part A.
- Part C: Surgery sub-trial: This part of the trial included any of the patients from Part A and Part B that during the course of the trial needed to undergo a major or minor surgical procedure requiring at least 7 days of daily FVIII treatment, including the day of surgery. Patients received a preoperative loading dose of turoctocog alfa immediately prior to the surgical procedure. On the day of surgery and until Day 7 (included) turoctocog alfa was dose adjusted aiming for a trough level above 0.50 IU/mL. Day 8 to last day of the surgical recovery period (if relevant) turoctocog alfa was dosed according to local guidelines.
Arm/Group | Total (Part A + Part B) | Part C | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 150 | 9 | 150
events
  All AEs | 222 | 3 | 225
  Severe AEs | 8 | 0 | 8
  Moderate AEs | 51 | 1 | 52
  Mild AEs | 163 | 2 | 165
  Serious AEs | 9 | 0 | 9
  Probably or Possibly Related | 17 | 0 | 17

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 188 days per subject.
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Arm/Group | All Subjects Treated With Turoctocog Alfa
Serious Adverse Events (participants affected / at risk) | 7/150
Other Adverse Events (participants affected / at risk) | 36/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated With Turoctocog Alfa (N=150)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated With Turoctocog Alfa (N=150)
Nasopharyngitis (Infections and infestations) | 12 (13)
Incorrect dose administered (Injury, poisoning and procedural complications) | 15 (19)
Headache (Nervous system disorders) | 14 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained during the conduct of this trial is considered confidential and can be used by Novo Nordisk for regulatory purposes and for the general development of the trial product. The information obtained during this trial may be made available to other physicians who are conducting other clinical trials with the trial product, if deemed necessary by Novo Nordisk.